CLINICAL TRIAL: NCT04690517
Title: Comparison of Tracheal Ultrasound With Capnography for Intubation Confirmation During CPR (Cardiopulmonary Resuscitation) Wearing PPE (Personnel Protective Equipment): A Prospective Comparative Study
Brief Title: Comparison of Tracheal Ultrasound With Capnography for Intubation Confirmation During CPR Wearing PPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-11-115
Record Dates: First submitted 2020-12-21; First posted 2020-12-30 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2020-12

CONDITIONS: Cardiopulmonary Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tracheal ultrasound (Other): The patients in cardiopulmonary arrest should be performed tracheal ultrasound when tube is passed through the trachea or esophagus.
  Interventions: Procedure: tracheal ultrasound

INTERVENTIONS:
Procedure: tracheal ultrasound — When checking tracheal ultrasound, several signs are used in judgements. Direct signs include reverberation artifact and double ring sign. Indirect sign means checking the bilateral lung sliding.

SUMMARY:
It is very important to ensure the tube placement in patients with cardiac arrest and unrecognized misplacement of endo-tracheal tube can lead to morbidity and mortality. In recent pandemic situations such as COVID-19 (Coronavirus disease-19), the number of cases of cardiopulmonary resuscitation with personal protective equipment (PPE) have increased. In those cases, existing methods such as auscultation and chest uprising have to be limited. Quantitative waveform capnography is recommended as the gold standard for confirming correct endotracheal tube placement in the 2010 American HeartAssociation (AHA) Guidelines for Cardiopulmonary resuscitation (CPR) and Emergency Cardiovascular Care (ECC), but it has some well-known limitations in cardiac arrest patients.

Ultrasonography is a non-invasive, real-time diagnostic tool commonly used during resuscitation. Especially, tracheal ultrasonography can be performed in real-time when the tube is passed through the trachea or esophagus. Previous prospective studies revealed that tracheal ultrasonography could feasibly and rapidly confirm tracheal intubation during emergency intubation.

There have already been several studies comparing the accuracy of tracheal ultrasound and capnography, but there was no study comparing the two tools under the constraints of PPE that is essential in pandemic situations as in this study. This study aimed to determine the accuracy of tracheal ultrasonography in assessing endotracheal tube position during CPR with PPE.

DETAILED DESCRIPTION:
When patients in cardiopulmonary arrest enter a emergency room (ER) or patients staying in a ER have a cardiopulmonary arrest, participants perform intubation and CPR. When it is judged as a high-risk group with a high probability of droplet infection, all participants in resuscitation team should wear personal protective equipment. Tracheal ultrasound and end-tidal carbon dioxide are used to confirm the placement of tube. The gold standard is the direct visualization using laryngoscope. The time it takes to confirm the placement of tube is also measured.

ELIGIBILITY:
Inclusion Criteria:

* 1. cardiopulmonary arrest patients receiving emergency intubation and CPR
* 2. patients judged to need to wear PPE according to the judgement of the clinician

Exclusion Criteria:

* 1. sign for "do not resuscitate (DNR)"
* 2. patients unable to perform tracheal ultrasound due to trauma of the site
* 3. patients unable to perform tracheal ultrasound due to oropharynx cancer
* 4. patients unable to perform tracheal ultrasound due to placement of tracheal cannula
* 5. patients not used tracheal ultrasound for checking tube placement

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-01-30 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Accuracy | during intubation procedure
  The gold standard is direct visualization using laryngoscopy. Tracheal ultrasound is performed regardless of whether it is in real-time or not.

CONTACTS AND LOCATIONS:
Overall Officials: Hee Yoon, Professor, Study Chair — Samsung medical center, Emergency department
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chou HC, Chong KM, Sim SS, Ma MH, Liu SH, Chen NC, Wu MC, Fu CM, Wang CH, Lee CC, Lien WC, Chen SC. Real-time tracheal ultrasonography for confirmation of endotracheal tube placement during cardiopulmonary resuscitation. Resuscitation. 2013 Dec;84(12):1708-12. doi: 10.1016/j.resuscitation.2013.06.018. Epub 2013 Jul 9. PMID 23851048